CLINICAL TRIAL: NCT03505476
Title: Optimizing the Previs Device for Prediction of Postoperative Ileus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jennifer Hrabe (Other)
Responsible Party: Sponsor-Investigator, Jennifer Hrabe, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201801808
Record Dates: First submitted 2018-04-11; First posted 2018-04-23 (Actual); Results first posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-02

CONDITIONS: Ileus
Keywords: Ileus; Abdominal surgery; Bowel obstruction; Postoperative Ileus
MeSH Terms: conditions — Ileus; Intestinal Obstruction

STUDY DESIGN:
Intervention Model Description: All subjects consented and enrolled will receive the same intervention. There is no control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Study Participants (Experimental): Device: Entac Medical device application Other: Patient Daily Assessment Other: Patient Discharge Assessment
  Interventions: Device: Entac Medical device application; Other: Patient Daily Assessment; Other: Patient Discharge Assessment

INTERVENTIONS:
Device: Entac Medical device application — Subjects will wear a 3-inch by 3-inch stethoscope device that adheres to the skin of the abdomen via FDA approved adhesive material. It will be applied either in the operating room at the completion of surgery or in the recovery room. The device will remain on the abdomen until discharge or for 10 days, whichever comes first.
Other: Patient Daily Assessment — The research team will ask questions of the subject regarding nausea, vomiting, passage of flatus, return of bowel function, and satisfaction with the device every day that the subject is hospitalized.
Other: Patient Discharge Assessment — The research team will ask questions of the subject regarding satisfaction or dissatisfaction with having the device placed and attached to their abdomen.

SUMMARY:
The research proposed in this study will develop a noninvasive prototype device that will capture intestinal sounds, process signals, and display predictive information in real-time at the point-of-care using algorithms already developed at this institution.

DETAILED DESCRIPTION:
Following major abdominal surgery, up to 30% of patients develop a poorly understood condition known as ileus. When ileus occurs, the bowels shut down and patients often develop abdominal dissension, nausea, vomiting, and even more serious complications. Because this condition does not develop until many days after surgery has been completed, clinicians do not know if they should begin allowing patients to eat or withhold nutrition until they show signs of bowel function such as passing gas or having bowel movements. Clinicians have different approaches but none are ideal: 1) feed all patients early and the ones that develop an ileus will have their diets reverse, suction tube placed in their stomach, and hopefully don't get develop more serious complications, or 2) don't feed patients until they pass gas or have a bowel movement, which delays nutrition and prolongs hospital stays for the 70% of patients who will not develop an ileus

Participants in this study will be asked to wear a 3-ounce device that adheres to the skin of the abdominal wall for 10 days. They will also be asked to answer questions each day of their hospital stay regarding how they have tolerated eating.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing elective intestinal resection surgery by the colorectal surgery service at UIHC.

Age 18 to 100.

Exclusion Criteria:

Allergies to any of the device components. Inability to have prototype device applied to their abdominal wall due to a condition (ie:fistulas, stomas, drains, etc).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Hrabe, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Participants
Started | 203
Completed | 75
Not Completed | 128
Not completed — Physician Decision | 18
Not completed — Device Malfunctioned | 101
Not completed — Data Corrupt | 6
Not completed — Device application insufficiant | 3

BASELINE CHARACTERISTICS:
Arm/Group | Study Participants
Number analyzed (Participants) | 203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 139
  >=65 years | 64
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108
  Male | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 197
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 195
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 203

OUTCOME MEASURES:

1. Primary Outcome: Device Sensitivity for Predicting Ileus.
Description: Calculate the sensitivity of the device to predict ileus, as defined by the number of patients with device-predicted ileus (true positive) as compared to the number both with device-predicted ileus and with ileus that the device did not predict (true positive + false negative).
Time Frame: Each patient's device's data was assessed at day 15.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Participants
Number analyzed (Participants) | 75
Participants
  Patients with Ileus whose device predicted ileus (true positive). | 12
  Patients with ileus whose device did not predict ileus (false negative). | 2
  Patients without ileus whose device predicted ileus (false positive). | 22
  Patients without ileus whose device did not predict ileus (true negative). | 39

2. Primary Outcome: Device Specificity for Predicting Ileus
Description: Calculate the specificity of the device to predict ileus, as defined by the number of patients where the device correctly predicted no ileus (true negative) as compared to the number both with device correctly predicting no ileus and device incorrectly predicting ileus (true negative plus false positive).
Time Frame: Each patient's device's data was assessed at day 15.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Participants
Number analyzed (Participants) | 75
Participants
  Patients with ileus whose device predicted ileus (true positive) | 12
  Patients with ileus whose device did not predict ileus (false negative) | 2
  Patients without ileus whose device predicted ileus (false positive) | 22
  Patients without ileus whose device did not predict ileus (true negative) | 39

3. Primary Outcome: Device Positive Predictive Value for Predicting Ileus
Description: Calculate the positive predictive value of the device to predict ileus, as defined by the number of patients with device-predicted ileus (true positive) as compared to the number both with device-predicted ileus and with device incorrectly predicting ileus (true positive plus false positive).
Time Frame: Each patient's device's data was assessed at day 15.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Participants
Number analyzed (Participants) | 75
Participants
  Patients with ileus whose device predicted ileus (true positive) | 12
  Patients with ileus whose device did not predict ileus (false negative) | 2
  Patients without ileus whose device predicted ileus (false positive) | 22
  Patients without ileus whose device did not predicted ileus (true negative) | 39

4. Primary Outcome: Device Negative Predictive Value for Predicting Ileus
Description: Calculate the negative predictive value of the device to predict ileus, as defined by the number of patients where the device correctly predicted no ileus (true negative) as compared to the number both with device correctly predicted no ileus and with ileus the device did not predict (true negative plus false negative).
Time Frame: Each patient's device's data was assessed at day 15.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Participants
Number analyzed (Participants) | 75
Participants
  Patients with ileus whose device predicted ileus (true positive) | 12
  Patients with ileus whose device did not predict ileus (false negative) | 2
  Patients without ileus whose device predicted ileus (false positive) | 22
  Patients without ileus whose device did not predicted ileus (true negative) | 39

ADVERSE EVENTS:
Time Frame: Adverse event data was collected on all subjects until their study participation is completed. (typically at or around 14 days)
Arm/Group | Study Participants
All-Cause Mortality (participants affected / at risk) | 0/203
Serious Adverse Events (participants affected / at risk) | 0/203
Other Adverse Events (participants affected / at risk) | 0/203

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/76/NCT03505476/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT03505476/SAP_001.pdf